CLINICAL TRIAL: NCT03579225
Title: Improving the Efficiency of the Digital Sleep Workflow Using MATRx Plus
Status: Completed | Type: Observational
Sponsor: Zephyr Sleep Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: ZCP201801
Record Dates: First submitted 2018-06-25; First posted 2018-07-06 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (1):
- MATRx plus test
  Interventions: Device: MATRx plus test

INTERVENTIONS:
Device: MATRx plus test — The MATRx plus is a home-based test that allows the healthcare provider to determine if a patient with obstructive sleep apnea will benefit from oral appliance therapy. Prior to the test, a dentist fits the patient with dental trays and measures the patient's comfortable jaw range of motion. The trays are connected to a mandibular positioner. During sleep, the device collects airflow from a nasal cannula and blood oxygen saturation from a pulse oximeter. These signals are used by the device software to control the mandibular positioner and protrude the mandible. During the test, the device moves the lower jaw within the patient's range of motion to predict if the patient is likely to benefit from oral appliance therapy and, if so, the appropriate amount of protrusion. Additional study nights may be required if the data from either of the first two nights are insufficient or if a more precise determination of the amount of jaw protrusion that provided a therapeutic benefit can be made.

SUMMARY:
Sleep apnea (OSA) is a condition in which the air passage in the throat closes or partly closes during sleep and repeatedly interrupts breathing. The standard treatment for sleep apnea is continuous positive airway pressure (CPAP), but it is not suitable for all patients. Another treatment is to use an oral appliance in your mouth when you sleep. The appliance covers the upper and lower teeth and pulls the lower jaw forward, opening the airway and allowing normal breathing.

Oral appliance treatment does not treat sleep apnea effectively in all patients. To identify patients for whom oral appliance therapy will work, Zephyr Sleep Technologies invented a device that tests various positions of the lower jaw from the comfort of your own home. The MATRx plus device is considered investigational since it has not been cleared by the U.S. FDA. During the MATRx plus test, the patient sleeps with a motorized positioner that moves the lower jaw. Jaw movement is automatically controlled by a computer, making the device a feedback controlled mandibular positioner.

The purpose of the study is to test the workflow of the MATRx plus feedback controlled mandibular positioner in its intended setting. The workflow includes recruitment into the study, the screening process, visits at the dentist, home sleep tests, and the decision made regarding oral appliance therapy based on the results of the sleep tests. The main objective is to determine the turnaround time of a MATRx plus test in a real-use dental setting.

DETAILED DESCRIPTION:
Sleep apnea (OSA) is a condition in which the air passage in the throat closes or partly closes during sleep and repeatedly interrupts breathing. The standard treatment of sleep apnea is continuous positive airway pressure (CPAP), but it is not suitable for all patients. Another treatment is to use an oral appliance in your mouth when you sleep. The appliance covers the upper and lower teeth and pulls the lower jaw forward, opening the airway and allowing normal breathing.

Oral appliance treatment does not treat sleep apnea effectively in all patients. To identify patients for whom oral appliance therapy will work, Zephyr Sleep Technologies has invented a remotely controlled device that tests various positions of the lower jaw. This commercially available device, MATRx, is a U.S. Food and Drug Administration (FDA)-cleared motorized positioner that is used in an overnight sleep study performed in the hospital or clinic.

During the test, temporary dental impression trays cover the upper and lower teeth. These are attached to a small motor that slowly and gently pulls the lower jaw forward under the control of a technician who determines when the best position is reached. Knowing the best position and the likelihood of therapy success allows the dentist to build an oral appliance with confidence.

To eliminate the need for an overnight in-hospital study, Zephyr Sleep Technologies has invented a new investigational device that allows us to decide if patients are likely to benefit from oral appliance therapy from the comfort of the patient's own home. An investigational device is one that is not cleared by the U.S. FDA. Like MATRx, the patient sleeps with a motorized positioner that moves the lower jaw. However, the new device (MATRx plus) is automatically controlled by a computer, rather than a sleep technician, making it a feedback controlled mandibular positioner.

We have previously carried out four research studies leading to the development of this feedback controlled mandibular positioner. The first study showed that the technician-controlled positioner was able to accurately identify patients who were suitable for oral appliance therapy. This study also identified the amount of jaw protrusion needed to provide therapeutic relief of the patients' sleep apnea. This trial resulted in the placement of the MATRx device on the market. The other three trials showed that the feedback-controlled software used by the new positioner was very accurate and was able to identify successful candidates in a home setting.

No serious or permanent problems or risks were identified in any of the research studies. Participants reported minor tooth and gum discomfort on the morning following the test and other minor issues, including excess saliva and being unable to sleep. Since other studies were designed to establish the safety and efficacy of the device, the purpose of the present research study is to collect data regarding the use of the device in its intended commercial setting, i.e., the dentist's office.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* suitable for oral appliance therapy
* ability to understand and provide informed consent
* ability and willingness to meet the required schedule

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study participants will be recruited from the Principal Investigator's population of patients.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-04-14 (Actual); Study Completion 2019-04-14 (Actual)

PRIMARY OUTCOMES:
Device turnaround time | 1 week
  Time from device deployment for MATRx plus test to device return (days).

CONTACTS AND LOCATIONS:
Locations (1):
- Raleigh Dental Arts, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No